CLINICAL TRIAL: NCT06596109
Title: Lifestyle Changes in Fatty Liver; Additive Effect of Honey Intake
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005163
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- honey intake and lifestyle changes (Experimental): Twenty fatty liver (non-alcoholic from) patients with obesity are included as 20 patients who will receive honey intake (orally, as a daily total dose of 2 g/kg, this dose will be divided to three equal subdoses, every dose will be administered before meal), low calorie diet, and treadmill walking (40 minutes per session, three times per week) for 12 weeks.
  Interventions: Behavioral: honey intake and lifestyle changes
- lifestyle changes (Active Comparator): Twenty fatty liver (non-alcoholic from) patients with obesity are included as 20 patients who will receive low calorie diet, and treadmill walking (40 minutes per session, three times per week) for 12 weeks.
  Interventions: Behavioral: lifestyle changes

INTERVENTIONS:
Behavioral: honey intake and lifestyle changes — Twenty fatty liver (non-alcoholic from) patients with obesity are included as 20 patients who will receive natural unprocessed honey intake (orally, as a daily total dose of 2 g/kg, this dose will be divided to three equal subdoses, every dose will be administered before meal), low calorie diet, and treadmill walking (40 minutes per session, three times per week) for 12 weeks.
  Arms: honey intake and lifestyle changes
Behavioral: lifestyle changes — Twenty fatty liver (non-alcoholic from) patients with obesity are included as 20 patients who will receive low calorie diet and treadmill walking (40 minutes per session, three times per week) for 12 weeks.
  Arms: lifestyle changes

SUMMARY:
honey is a natural functional food used in control cardiovascular risk factors but its effect on fatty liver is not investigated

DETAILED DESCRIPTION:
Forty fatty liver (non-alcoholic from) patients with obesity are included to be divided into group 1 who will contain 20 patients who will receive honey intake (orally, as a daily total dose of 2 g/kg, this dose will be divided to three equal subdoses, every dose will be administered before meal), low calorie diet, and treadmill walking (40 minutes per session, three times per week) for 12 weeks. Group 2 who will contain 20 patients who will receive low calorie diet, and treadmill walking (40 minutes per session, three times per week) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* fatty liver (non alcoholic form)
* both sexes included
* obese subjects (class I)

Exclusion Criteria:

* cardiac insult
* respiratory insult
* renal insult
* lower limb insult

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
High density lipoprotein | it will be assessed after 12 weeks
  it will be measured in serum

SECONDARY OUTCOMES:
triglycerides | it will be assessed after 12 weeks
  it will be measured in serum
cholesterol | it will be assessed after 12 weeks
  it will be measured in serum
low density lipoprotein | it will be assessed after 12 weeks
  it will be measured in serum
alanine transamianse | it will be assessed after 12 weeks
  it will be measured in serum
aspartate transamianse | it will be assessed after 12 weeks
  it will be measured in serum
fasting blood glucose | it will be measured after 12 weeks
  it will be measured in serum
body mass index | it will be measured after 12 weeks
  it will be measured on empty stomach
waist circumference | it will be measured after 12 weeks
  it will be measured on empty stomach

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt